CLINICAL TRIAL: NCT06314607
Title: Genetic and Molecular Characterization of Nervous System Lesions
Acronym: ONCONEUROTEK 2
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220498
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Brain Tumor; Brain Lesion (General)
Keywords: Brain tumor; Cerebral Lesions
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Constitutional DNA analysis covers :
  * the study of polymorphisms (SNPs) common in the general population, enabling GWAS (Genome Wide Association Studies) but not the detection of genetic anomalies.
  * analysis of coding sequences (whole exome/genome sequencing), which may be necessary in the following situations:
    * in order to interpret validly the results obtained by whole exome/genome sequencing of tumor DNA
    * in cases of suspected genetic predisposition to the development of brain tumors or lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Patients already included in the first ONCONEUROTEK (retrospective) study and followed up in the participating center : at their next hospitalization or consultation at Pitié Salpêtrière, they will be given an information note and a consent form (NIFC) informing them of the ONCONEUROTEK 2 study.
  (This population concerns all patients in the relevant departments with a last news date < 2 years)
  Interventions: Genetic: Prospective Biological Collection; Genetic: Retrospective Biological Collection
- Group 2: Patients included prospectively : Patients who may be included in this study will be informed of its objectives and procedures by the doctor in charge of their follow-up, during a consultation visit or routine hospitalization, by means of an information note.
  (This population concerns around 1,000 patients per year, i.e. around 10,000 patients over 10 years)
  Interventions: Genetic: Prospective Biological Collection; Genetic: Retrospective Biological Collection
- Group 3: This group concerns patients already included in the ONCONEUROTEK study (retrospective) but not currently being followed at the Pitié Salpêtrière hospital. Specifically, patients who are known to the investigators to still be alive. In this case, an information note and a non-opposition form (NINO) will be sent to them by mail to :
  * inform them of the regulatory update under the Loi Jardé and the RGPD
  * and collect their non-opposition to the re-use of their data and samples.
  * If no reply is received within one month, the patient will be deemed not to have objected to the re-use of his or her data and samples in the ONCONEUROTEK 2 study.
  (This population concerns all patients in the relevant departments with a last news date > 2 years)
  Interventions: Genetic: Retrospective Biological Collection

INTERVENTIONS:
Genetic: Prospective Biological Collection — All samples that can be collected at each visit :
  * Saliva sampling (added by the research)
  * Collection of 2 to 4 additional tubes of blood (maximum 56mL) (added by the research if blood sampling in routine care)
  * Urine and stool samples (added by the research)
  * CSF sample residues (added by the research if lumbar punction in routine care)
  * Lesion sample residues and surgical waste fragments (added by the research if surgery in routine care)
  Groups: Group 1; Group 2
Genetic: Retrospective Biological Collection — Requalification of all biological samples obtained as part of ONCONEUROTEK research, with patient consent (blood, saliva, urine, Stool, CSF, lesion sample and surgical waste fragments)

SUMMARY:
Primary and secondary brain tumors, the leading cause of death from cancer before the age of 35, represent a complex and heterogeneous group of pathologies with a generally poor prognosis. Knowledge of these tumors has made enormous strides thanks to access to biological samples, leading to a much more robust, reliable and precise histo-pronostic classification, but also, increasingly, to the identification of theranostic targets.

Despite these advances, there is a real need to refine diagnostic and prognostic classification, identify the biological mechanisms involved in the formation and progression of these pathologies, develop new targeted strategies, and devise minimally invasive follow-up methods (liquid biopsies).

In addition, certain non-tumoral brain lesions (e.g. malformations) can be similarly classified according to their molecular and mutational profile.

This project aims to make a decisive contribution to these objectives.

DETAILED DESCRIPTION:
Over the past 15 years, knowledge of these tumors has increased exponentially, thanks to the genomic revolution (high-throughput sequencing, methylome analysis), which has improved their classification, defining homogeneous prognostic, predictive and even theranostic groups (BRAF, FGFR, NTRK). This knowledge has only progressed thanks to access to tumor samples, but also to constitutional DNA and liquid biopsies.

The histo-pronostic classification of these tumors is constantly evolving, as evidenced by the new WHO 2021 version, which integrates more and more molecular markers for diagnosis (in which the team participated), and considerably modifies nosological frameworks. This process began with the 2007 classification, which was purely morphological and particularly unsatisfactory, with over 30% inter-observer diagnostic discordance, and the 2016 version has considerably clarified the classification of grade 2 and 3 gliomas, by integrating biomarkers that are now unavoidable, such as 1p19q codeletion and IDH1 and IDH2 mutation: however, it has taken several years for these markers to be routinely performed and managed. The extremely rapid evolution of diagnostic criteria is illustrated by the c-impact now initiative, which has regularly revisited the classification of primary brain tumours, and gliomas in particular, in the light of the most recent publications, and on which the 2021 classification is based: however, certain data are still fragile and criticized because they are based on limited series (for example, the definition of grade 2 gliomas, reclassified as "molecular glioblastomas".

Glioblastoma and other diffuse gliomas are incurable, lethal diseases that are resistant to conventional treatments (radiotherapy, chemotherapy). Compared with other cancers, the number of effective treatments and therefore treatment lines available is limited. The longitudinal study of these diseases is essential to understanding the mechanisms of resistance to treatment and identifying new vulnerabilities. Our team actively contributes to this research, for which tumor samples at initial diagnosis, but also at recurrence and possibly post-mortem are invaluable.

Given its strengths, our team can now make a decisive contribution to improving diagnosis and prediction in the management of primary brain tumors.

First and foremost, the team represents Europe's leading center for the management of glioma patients. Between 10% and 15% of patients with primary brain tumors in France are treated in Neuro-oncology at La Salpêtrière.

Beyond the diagnostic aspect, high-throughput sequencing techniques have made it possible to identify anomalies that can be used in oncology. However, these are still rarely detected in gliomas. Only a very limited number of markers, included in the WHO2016 classification, which we helped to identify, are now part of the "standard" management of these patients. The rest are part of research. However, we have recently shown that a broader search for actionable abnormalities carried out in specific studies, has enabled patients to benefit from personalized therapies with a real gain in survival, but access is still restricted via the Seqoia program, to a small number of patients.

In conclusion, there is a real need to refine diagnostic and prognostic classification, identify new targeted strategies, and develop minimally invasive follow-up methods (liquid biopsies).

Some lesions, however, are not tumoral in nature, but rather malformative, such as cerebral dysplasia or vascular malformations. Interestingly, somatic mutations are also found at the origin of these lesions, making it possible to classify them, and above all to propose treatments targeting these alterations. As these non-tumoral lesions are subject to a diagnostic and sometimes therapeutic strategy similar to tumors, and as our team has developed real expertise in this field, and above all as it is not always possible to distinguish, pre-operatively, between a malformative lesion and a tumor, we have broadened the search, and retain the term "lesion" in the patient information and consent form.

ELIGIBILITY:
Inclusion Criteria:

* Any patient operated on for a brain lesion (e.g. tumors: glioma, LCPSNC, meningioma, or rare tumor) and/or followed up for one of these pathologies.
* Age ≥ 18 years
* Consent or non-opposition of the patient or his/her legal representative (guardian) to participate in the study.

Exclusion Criteria: NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with brain lesions, including pregnant women (e.g. tumors: patient with glioma, but also with primary brain lymphoma, meningioma, or primary brain tumor of a rare subtype, secondary tumor).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Study the clinical markers with the evolution of brain lesions. | 10 years
  Study of patients' disease-related data in their medical records
Study the biological markers with the evolution of brain lesions. | 10 years
  Study blood, saliva, urine, stool and CSF samples
Study the anatomopathological markers with the evolution of brain lesions. | 10 years
  Study of cerebral lesion tissues

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Neurochirurgie - Hôpital de la Pitié Salpêtrière, Paris
  - Service de Neurologie 2 -Hôpital de la Pitié Salpêtrière, Paris
  - Service de Radiothérapie - Hôpital de la Pittié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided